CLINICAL TRIAL: NCT01353729
Title: A Phase I, Randomized, Placebo-Controlled, Four-Way Crossover Study to Evaluate the Effect of Intravenous (IV) Zanamivir on Cardiac Conduction as Assessed by 12-lead Electrocardiogram (ECG) With Moxifloxacin as a Positive Control in Healthy Volunteers
Brief Title: A Study to Evaluate the Effect of Intravenous Zanamivir on Cardiac Conduction in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 114346
Record Dates: First submitted 2011-05-12; First posted 2011-05-16 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Influenza, Human
Keywords: 12-lead ECG; cardiac repolarization; QTc; influenza; GR121167; zanamivir
MeSH Terms: conditions — Influenza, Human | interventions — Zanamivir; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment A (Experimental): Treatment A will include combination of zanamivir 600 mg IV plus placebo for moxifloxacin
  Interventions: Drug: 600 mg zanamivir + moxifloxacin placebo
- Treatment B (Experimental): Treatment A will include combination of zanamivir 1200 mg IV plus placebo for moxifloxacin
  Interventions: Drug: 1200 mg zanamivir + moxifloxacin placebo
- Treatment C (Experimental): Treatment C will include zanamivir placebo plus placebo for moxifloxacin
  Interventions: Drug: zanamivir placebo + moxifloxacin placebo
- Treatment D (Experimental): Treatment D will include moxifloxacin plus zanamivir placebo
  Interventions: Drug: zanamivir placebo + 400 mg moxifloxacin

INTERVENTIONS:
Drug: 600 mg zanamivir + moxifloxacin placebo — zanamivir 600 mg IV over 30 min x 1 dose + moxifloxacin placebo administered orally x 1 dose
  Arms: Treatment A
Drug: 1200 mg zanamivir + moxifloxacin placebo — zanamivir 1200 mg IV over 30 min x 1 dose + moxifloxacin placebo administered orally x 1 dose
  Arms: Treatment B
Drug: zanamivir placebo + moxifloxacin placebo — zanamivir placebo IV over 30 min x 1 dose + moxifloxacin placebo administered orally x 1 dose
  Arms: Treatment C
Drug: zanamivir placebo + 400 mg moxifloxacin — moxifloxacin 400 mg administered orally x 1 dose + zanamivir placebo IV over 30 min x 1 dose
  Arms: Treatment D

SUMMARY:
Approximately 40 healthy subjects will be enrolled. Each subject will participate in the study for approximately 9 weeks. There will be four treatment sequences with a 5-7 day washout between treatments. Subjects will be admitted to the clinical unit on Day-1 of each dosing period and will remain in the unit until Day 2. Each subject will receive a single dose of each of the four treatments on Day 1 of each treatment period in a randomized fashion. Subjects will be discharged from the clinical research unit after the completion of all assessments on Day 2 of each period and return approximately 5-7 days later for the next dose period. Serial pharmacokinetic samples will be collected for up to 24 hours following each treatment.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring.
* Male or female between 18 and 55 years of age inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea or of child-bearing potential and agrees to use one of the contraception methods listed in the protocol.
* Body weight greater than or equal to 50 kg for men and greater than or equal to 45 kg for women and BMI within the range 18.5-31.0 kg/m2 (inclusive).
* AST, ALT, alkaline phosphatase and bilirubin less than or equal to 1.5xULN (isolated bilirubin >1.5x upper limit of normal (ULN) is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Capable of giving written informed consent, which includes agreement to comply with the requirements and restrictions listed in the consent form

Exclusion Criteria:

* The subject has a positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* History of sensitivity to any of the study medications, or components thereof, or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* A history of sensitivity to heparin or heparin-induced thrombocytopenia should not be enrolled.
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >14 drinks/week for men or >7 drinks/week for women.
* Has a history or regular use of tobacco- or nicotine-containing products within 3 months prior to screening.
* Pregnant females as determined by positive serum or urine human chorionic gonadotrophin (hCG) test at screening or prior to dosing.
* Lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subjects with a pre-existing condition interfering with normal gastrointestinal anatomy or motility, hepatic and/or renal function, that could interfere with the absorption, metabolism, and/or excretion of the study drugs. Subjects with a history of cholecystectomy, inflammatory bowel disease or pancreatitis should be excluded. Subjects with active peptic ulcer disease or a history of upper gastrointestinal bleeding
* A creatinine clearance less than 80mL/min as determined by Cockcroft-Gault equation.
* History/evidence of clinically significant pulmonary disease, renal or hepatobiliary diseases. Subjects with a history of nephrolithiasis will be excluded.
* A positive pre-study Human immunodeficiency virus (HIV) antibody test, a positive Hepatitis B surface antigen or Hepatitis C antibody result within 3 months of screening.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Subjects with a hemoglobin <11 g/dL. A single repeat is allowed for eligibility determination.
* The subject's systolic blood pressure is outside the range of 90-140mmHg, or diastolic blood pressure is outside the range of 45-90mmHg or heart rate is outside the range of 45-100bpm for female subjects or 45-100 bpm for male subjects.
* Exclusion criteria for screening ECG (a single repeat is allowed for eligibility determination) per protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2011-05-19 (Actual); Primary Completion 2011-08-02 (Actual); Study Completion 2011-08-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in QTcF for zanamivir | 9 weeks

SECONDARY OUTCOMES:
Change from baseline in QTcB | 9 weeks
Change from baseline in QTci | 9 weeks
Change from baseline in QT | 9 weeks
Change from baseline in Heart Rate | 9 weeks
Pharmacokinetic parameters of Area under the concentration-time curve from time zero (pre-dose) to time of last quantifiable concentration from serum zanamivir concentration-time data | 9 weeks
Pharmacokinetic parameters of Area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time from serum zanamivir concentration-time data | 9 weeks
Pharmacokinetic parameters of maximum observed concentration from serum zanamivir concentration-time data | 9 weeks
Pharmacokinetic parameters of time of occurrence of cmax from serum zanamivir concentration-time data | 9 weeks
Pharmacokinetic parameters of systemic clearance of parent drug from serum zanamivir concentration-time data | 9 weeks
Pharmacokinetic parameters of volume of distribution in terminal phase from serum zanamivir concentration-time data | 9 weeks
Pharmacokinetic parameters of terminal phase half-life from serum zanamivir concentration-time data | 9 weeks
Pharmacokinetic parameters of Area under the concentration-time curve from time zero (pre-dose) to time of last quantifiable concentration (if needed) from plasma moxifloxacin concentration-time data | 9 weeks
Pharmacokinetic parameters of area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time (if needed) from plasma moxifloxacin concentration-time data | 9 weeks
Pharmacokinetic parameters of maximum observed concentration (if needed) from plasma moxifloxacin concentration-time data | 9 weeks
Pharmacokinetic parameters of time of occurrence of cmax (if needed) from plasma moxifloxacin concentration-time data | 9 weeks
Pharmacokinetic parameters of systemic clearance of parent drug (if needed) from plasma moxifloxacin concentration-time data | 9 weeks
Pharmacokinetic parameters of volume of distribution in terminal phase (if needed) from plasma moxifloxacin concentration-time data | 9 weeks
Pharmacokinetic parameters of terminal phase half-life (if needed) from plasm moxifloxacin concentration-time data | 9 weeks
Safety and tolerability of zanamivir as assessed by change from baseline in 12-lead Electrocardiograms (ECG) | 9 weeks
Safety and tolerability of zanamivir as assessed by change from baseline in blood pressure and heart rate | 9 weeks
Safety and tolerability of zanamivir as assessed by change from baseline in the collection of adverse events | 9 weeks
Safety and tolerability of zanamivir as assessed by change from baseline in toxicity grading of clinical laboratory tests | 9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Lou Y, Gan J, Peppercorn A, Gould E, Weller S, Piscitelli SC, Patel P. Effect of intravenous zanamivir on cardiac repolarization. Pharmacotherapy. 2013 Jul;33(7):701-9. doi: 10.1002/phar.1261. Epub 2013 Apr 3. PMID 23553534
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 114346 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/114346?search=study&search_terms=114346#rs
- Available data/document: Annotated Case Report Form: 114346 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114346 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 114346 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114346 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114346 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114346 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114346 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register